CLINICAL TRIAL: NCT06276920
Title: Comparison of Elbow Joint Position Sense in Healthy Individuals in Open and Closed Kinetic Positions
Brief Title: Evaluation of Joint Position Sense in Healthy Individuals
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gülfem Ezgi ÖZALTIN, PhD, physiotherapist, Principal Investigator, Inonu University
Other Study IDs: 2024/5554(1)
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Proprioception
Keywords: Proprioception; Joint Position Sense; healthy individuals; Open Kinetic Position; Closed Kinetic Position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It was aimed to measure the elbow joint position sense in healthy individuals in the case of a closed kinetic chain and to compare it with the measurement made in the case of an open kinetic chain.

DETAILED DESCRIPTION:
The study was designed as a non-invasive, cross-sectional study. The population of this research will consist of healthy individuals. Joint position sense will be measured in open kinetic chain and closed kinetic chain via universal goniometer . Each angle position will be repeated 3 times with the elbow in 45, 60, 75 degree flexion angle positions and the average will be calculated. Measurements will be evaluated simultaneously but independently with the 2 different evaluators. Measurements will be repeated after 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being healthy
* Agreeing to participate in the study

Exclusion Criteria:

* Those who have had upper extremity surgery within the last year
* Those with neurological, orthopedic, rheumatic or cardiovascular problems affecting the neck, shoulder, elbow, hand and wrist
* Those with central and peripheral nervous system involvement Having pain anywhere in the body

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Joint position sense measurement with universal goniometer in close kinetic chain | 3 days
  In the closed kinetic chain, measurements are made at different starting positions.
Joint position sense measurement with universal goniometer in open kinetic chain | 3 days
  In the open kinetic chain, joint position sense is measured as the subject's ability to actively reproduce the passively placed position of the forearm relative to the upper arm.

CONTACTS AND LOCATIONS:
Overall Officials: gulfem ezgi ozaltin, PhD, Principal Investigator — Inonu University; Dilan Demirtaş Karaoba, PhD, Study Chair — Inonu University; Havva Adli, Study Chair — Inonu University; burcu talu, Study Chair — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No